CLINICAL TRIAL: NCT06989424
Title: Visualization of the Colon Through Use of the Magnetic Flexible Endoscope (MFE) in Participants With Inflammatory Bowel Disease (IBD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Keith Obstein, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: MFEIBD_241894; 5R01EB018992-08 (NIH)
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Bowel Disease (IBD); Colonoscopy
Keywords: Colonoscopy; Colon; Robotic; Magnetic; Endoscopy; Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (SOC) colonoscopy followed by Magnetic Flexible Endoscope (MFE) (Experimental): Patients in this group will have their SOC colonoscopy for IBD/colorectal cancer screening completed with a legacy colonoscope followed by colonoscopy with the MFE.
  Interventions: Device: Magnetic Flexible Endoscope (MFE)
- Colonoscopy with Magnetic Flexible Endoscope (MFE) followed by Standard of Care (SOC) colonoscopy (Experimental): Patients in this group will have colonoscopy with the MFE followed by the legacy colonoscope for standard of care IBD/colorectal cancer screening.
  Interventions: Device: Magnetic Flexible Endoscope (MFE)

INTERVENTIONS:
Device: Magnetic Flexible Endoscope (MFE) — The Magnetic Flexible Endoscope (MFE) is a single-use endoscope intended to integrate with other commercially available devices for visualization of the human colon in order to eliminate the need for passage of the much stiffer, non-intuitive, risk prone standard colonoscope. The MFE will be introduced into the colon and traverse from the rectum to the cecum.

SUMMARY:
In this study, the investigators will test the ability of the Magnetic Flexible Endoscope (MFE) to travel through the colon of people with Inflammatory Bowel Disease (IBD). The MFE is a device made of ultra-flexible tubing that contains a camera, light, and magnet at the tip. The tip of the tube is about the size of a penny. The magnet inside the tip allows the MFE to be moved through the colon by a second magnet attached to a robotic arm that is outside the body. The purpose of this study is to see how the MFE travels through the colon of IBD patients and if it is tolerable.

DETAILED DESCRIPTION:
Colonoscopy is the gold standard for making the diagnosis, following clinical response, establishing prognosis, and creation of management plans for patients with Inflammatory Bowel Disease (IBD). While colonoscopy is a relatively safe procedure, there are several limitations due to the unintuitive drive mechanism and mechanical design of current conventional colonoscopes. Additionally, for patients with IBD, the procedure is associated with a higher lifetime risk of adverse event due to increased frequency of examination-more than a 6-fold increased risk when compared to their non-IBD counterparts.

For these reasons, our team has developed a novel, highly compliant, Magnetic Flexible Endoscope (MFE) with the functionality of a conventional colonoscope (i.e. camera, therapeutic channel, irrigation, insufflation, illumination, lens cleaning). The MFE is driven by magnetic coupling of the endoscope head that contains an internal permanent magnet and a robotic arm that holds an external permanent magnet. This enables a "front-pull" actuation mechanism to eliminate the need for pushing a semi-rigid insertion tube for advancement. The forward drive mechanism thus prevents buckling of the insertion tube and avoids looping/colon wall stress. This reduces the risk of perforation and pain during the procedure to allow for less (if any) procedural sedation.

The Magnetic Flexible Endoscope (MFE) is a single-use endoscope intended to integrate with other commercially available devices for the visualization of a human colon in order to eliminate the need for passage of the much stiffer, non-intuitive, risk prone standard colonoscope. This study builds on the successful completion of the first-in-human feasibility study that demonstrated safety and tolerability in healthy patients who were already scheduled for their routine standard-of-care screening colonoscopy. In this secondary study, the MFE device will be inserted into the rectum via the anus and navigated through the colon to the cecum, using magnetic manipulation, in patients with stable, non-active, Inflammatory Bowel Disease (IBD) who are due for their IBD/colorectal cancer surveillance/screening colonoscopy exams.

The investigators plan to assess safety and tolerability of MFE navigation in the colon from the rectum to the cecum in patients with stable non-active IBD who are due for their IBD/Colorectal Cancer surveillance/screening colonoscopy exams. This will be a parallel study design in which three of six patients will have standard of care colonoscopy completed with monitored anesthesia care (MAC) first followed by MFE and three of six patients will undergo unsedated MFE first followed by standard of care colonoscopy completed with MAC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 70 years of age
* Able to provide written informed consent
* American Society of Anesthesiologists (ASA) class < 3
* No significant medical problems
* Abdominal circumference < 96 cm
* Stable, non-flaring inflammatory bowel disease (e.g. Ulcerative Colitis and Crohn's Disease)

Exclusion Criteria:

* Patients who do not meet inclusion criteria
* Patients who are unable or unwilling to provide informed consent
* Magnetic implants and wearable devices (such as insulin pumps)
* Females who are pregnant. As part of routine pre-operative care, all females of childbearing potential will undergo either urine or blood pregnancy testing.
* Cancer positive subjects or any patients currently undergoing any treatment or therapy to treat, cure, or mitigate cancer.
* Symptoms consistent with coronavirus (COVID-19) --- pyrexia, new persistent cough, or anosmia --- or a positive coronavirus (COVID-19) polymerase chain reaction (PCR) swab result
* Previous incomplete or failed colonoscopy
* Colonic resection
* Severe diverticulosis
* Known or suspected colonic stricture
* Previous radiation therapy to the abdomen or pelvis
* Actively flaring inflammatory bowel condition (e.g. active flare of IBD or diverticulitis)
* Known or suspected bowel obstruction
* Presence of ascites
* Participants taking anticoagulant medications or antiplatelet therapy (excluding aspirin) within the last 3 days
* Known coagulation disorder (INR ≥ 1.5 or platelets < 150 x 109)
* Known to have phenylketonuria or Glucose-6-Phosphate-Dehydrogenase (G6PD) deficiency
* Abdominal surgery within the last 6 months
* Drug or alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility to intubate the cecum (yes/no) | Day 1
  Ability to feasibly enter the cecum of the colon. Will be confirmed per standard endoscopic practice of visualizing and photo documenting at least 2 of the 3 common cecum landmarks (ileocecal valve, triradiate fold, appendiceal orifice).

SECONDARY OUTCOMES:
Mucosal visibility | Day 1
  Operator assessed score, the Colon Visualization Index, will be used. Scale ranges from 0 (poor) to 4 (excellent)
Patient tolerance | Day 1
  Pain perception will be assessed with a validated pain score (Wong-Baker FACES Pain Rating Scale) with 0 be no hurt to 10 hurts worst during a post-study structured interview.
Endoscopist experience | Day 1
  Usability of the platform in terms of task load for the endoscopist will be assessed using the standardized validated National Aeronautics and Space Administration (NASA) Task Load Index (TLX) based on a multidimensional construct of six sub-scales: mental demand, physical demand, temporal demand, performance, effort, and frustration level. The sub-scales range from 0 (very low) to 100 (very high): the exception is the sub-scale of performance, where 0 is perfect and 100 is failure.

CONTACTS AND LOCATIONS:
Overall Officials: Keith L Obstein, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT06989424/ICF_000.pdf